CLINICAL TRIAL: NCT07138456
Title: Clinical Severity of Dental Fluorosis and Associated Risk Factors Among a Group of Children in a Rural Region, Dendera Center in Egypt: A Cross-Sectional Study
Brief Title: Clinical Severity of Dental Fluorosis and Associated Risk Factors Among a Group of Children in Rural Region, Dendera Center in Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Gihad Mohamed Abdelraheem Abdelmajeed, Gihad Mohamed Abdelraheem Abdelmajeed, Cairo University
Other Study IDs: prevalence and severity of DF
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Dental Fluorosis
Keywords: prevalence, clinical severity and risk factors of dental fluorosis in a rural area in Egypt
MeSH Terms: conditions — Fluorosis, Dental

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of our observational study is evaluation of the clinical severity of dental fluorosis and associated risk factors among a group of children (8-12 years old) in a rural region, Dendera center, Egypt.

The main question it aims to answer is:

What is the clinical severity of dental fluorosis and associated risk factors among a group of children (8-12 years old) in a rural region, Dendera center, Egypt?

DETAILED DESCRIPTION:
Fluoride has a dual impact, it can be beneficial for dental health when consumed at optimal levels, but excessive intake can lead to a condition known as dental fluorosis (DF).

Dental fluorosis, which is particularly common among children and young individuals, is a developmental enamel defect caused by excessive fluoride exposure during the critical stages of tooth formation. This condition affects both the appearance and structure of the enamel.

The severity of dental fluorosis depends on various factors, including fluoride concentration in drinking water, daily intake, duration of exposure, and climatic conditions.

Epidemiological studies indicate that fluorosis can affect individuals across different age groups, with cases ranging from mild dental fluorosis to severe skeletal fluorosis. Children are particularly vulnerable to its harmful effects, which are often irreversible.

In rural areas, groundwater serves as the primary source of drinking water due to limited access to treated water supplies.

This dependence on groundwater increases the risk of prolonged fluoride exposure, particularly among children, whose developing teeth are more susceptible to fluorosis.

While several studies have documented the prevalence of dental fluorosis globally, there is a lack of data on its prevalence in rural areas of Upper Egypt, where groundwater is a key water source.

This knowledge gap highlights the need for localized research to assess the extent of the issue and develop targeted interventions.

Therefore, a cross-sectional study will be conducted to determine the prevalence and severity of dental fluorosis and identify associated risk factors among children in a rural area of the Dendera district, Qena governorate, Upper Egypt.

ELIGIBILITY:
Inclusion criteria:

* Children age range from 8 to 12 years.
* Children have lived in the area of the study since birth.
* Teeth to be examined should not be covered with fillings or braces.

Exclusion criteria:

* Parents or children who refuse to participate in the study.
* Ethical consideration.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Thy should be children with age range from 8 to 12 years, who have lived in the area of study since birth.
  the teeth to be examined should be clean and not covered with fillings or braces.
  the parents and children should accept to participate in the study and the parents should sign a consent according to ethical consideration.
Sampling Method: Non-Probability Sample
Enrollment: 231 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Clinically evident dental fluorosis in permanent incisors (prevalence) | Baseline (during the initial clinical examination of the child)
  Clinical examination (using a probe and mouth mirror in bright daily life, using ICMR index which have the following scores 0: no fluorosis /1: mild fluorosis _ 2: moderate fluorosis / 3: severe fluorosis)

SECONDARY OUTCOMES:
Clinically evident dental fluorosis in all permanent teeth present other than permanent incisors (prevalence) | Baseline (during the initial clinical examination of the child)
  Clinical examination (using a probe and mouth mirror in bright daily life, using ICMR index which have the following scores 0: no fluorosis /1: mild fluorosis _ 2: moderate fluorosis / 3: severe fluorosis)
Risk factors of dental fluorosis | baseline (upon enrollment, after parents complete the questionnaire)
  Multiple choice questions (questionnaire answered by the children's parents with multiple choice questions).
Severity of dental fluorosis | Baseline (during the initial clinical examination of the child)
  Scoring (0-3) according to Indian Council of Medical Research (ICMR) index which have the following scores 0: no fluorosis /1: mild fluorosis _ 2: moderate fluorosis / 3: severe fluorosis.

CONTACTS AND LOCATIONS:
Overall Officials: sarah A Mahmoud, PhD, Study Director — Cairo University
Locations (1):
- Dendera region, Cairo, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No